CLINICAL TRIAL: NCT00494104
Title: Prevention of Vitamin D Deficiency in Breastfed Infants
Brief Title: Prevention of Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD048870 (NIH); R01HD048870 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2006-09

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D deficiency; breastfed infant; northern latitude; infant; breastfed; winter; vitamin D status
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 200 IU/day Vitamin D (Active Comparator): 200 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D drops, 200 or 400 or 600 IU/day or 800 IU/day
- 400 IU/day Vitamin D (Experimental): 400 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D drops, 200 or 400 or 600 IU/day or 800 IU/day
- 600 IU/day Vitamin D (Experimental): 600 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D drops, 200 or 400 or 600 IU/day or 800 IU/day
- 800 IU/day Vitamin D (Experimental): 800 IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D drops, 200 or 400 or 600 IU/day or 800 IU/day

INTERVENTIONS:
Dietary Supplement: Vitamin D drops, 200 or 400 or 600 IU/day or 800 IU/day — Infants receive daily 0.5 ml of code labeled supplement

SUMMARY:
Breastfed infants living in a northern location (41 degrees N) are at high risk of vitamin D deficiency during winter. This trial is designed to determine how much supplemental vitamin D breastfed infants need to receive in order to remain free of vitamin D deficiency

DETAILED DESCRIPTION:
It is increasingly being recognized that infants and children living at northern latitudes are at risk of vitamin D deficiency, especially if their skin is darkly pigmented. The study by the PI (Pediatrics 2006;118:603) was the first to demonstrate that infants with light skin pigmentation living at 41 degrees north are at risk of vitamin D deficiency. During winter (December - April) a full 78% of infants were vitamin D deficient if they did not receive vitamin D from an external source. Very few breastfed babies are currently receiving supplemental vitamin D. The recommended dose is 200 IU/day. However, there are questions about the adequacy of this dose of vitamin D for the prevention of vitamin D deficiency. The present trial is designed to determine whether a dose of 200 IU/day is effective or whether doses of 400 IU/day, 600 IU/day or 800 IU/day are required to prevent vitamin D deficiency reliably.

The trial is a randomized, prospective double-blind trial in which breastfed infants will receive 200 IU/day or 400 IU/day or 600 IU/day or 800 IU/day from 1 to 9 months of age. There will not be a placebo control group. Infants will be followed through 12 months of age. Normal term infants (birth weight >2500 g) who are born in June through November will be enrolled and randomized at 1 month of age. They will visit the study center at monthly intervals and will have capillary blood drawn at select ages. At 2 months and again in March or April whole body mineral content will be determined by DEXA. Infants will not be permitted to receive formula until 9 months of age. They may receive complementary foods beginning at 4 months of age. Vitamin D supplements will be weighed before dispensing and again when the empty and half-empty containers are returned. Study endpoints will be blood parameters and bone mineral content determined at the end of winter, i.e., between March and May 15. Blood parameters include 25-OHD, parathyroid hormone, calcium, alkaline phosphatase, osteocalcin, N-telopeptide, ferritin and transferrin receptor. 180 infants will be enrolled at 1 month of age in the expectation that 48 per group will complete the trial to at least 9 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Term infant
* No major congenital malformations
* Less than one month old
* Breastfed, no other foods

Exclusion Criteria:

* Formula feeding
* Premature birth

Ages: 3 Weeks to 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 398 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of 25-hydroxyvitamin D, parathyroid hormone, alkaline phosphatase | end of winter

SECONDARY OUTCOMES:
whole body mineral content by DEXA | end of winter

CONTACTS AND LOCATIONS:
Overall Officials: Ekhard Ziegler, MD, Principal Investigator — University of Iowa
Locations (1):
- MTF, 2501 Crosspark Rd, Coralville, Iowa, United States

REFERENCES:
- [Derived] Ziegler EE, Nelson SE, Jeter JM. Vitamin D supplementation of breastfed infants: a randomized dose-response trial. Pediatr Res. 2014 Aug;76(2):177-83. doi: 10.1038/pr.2014.76. Epub 2014 May 23. PMID 24858141